CLINICAL TRIAL: NCT07022119
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Dose Extension Study Evaluating the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of VX-407 in Healthy Subjects
Brief Title: A Phase 1 Study Evaluating Safety, Tolerability, and Pharmacokinetics of VX-407 in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX24-407-002
Record Dates: First submitted 2025-06-06; First posted 2025-06-15 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease (ADPKD)
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: Single Ascending Dose (Experimental): Participants will be randomized to receive a single dose of VX-407.
  Interventions: Drug: VX-407
- Placebo Part A (Placebo Comparator): Participants will be randomized to receive placebo matched to VX-407.
  Interventions: Drug: Placebo
- Part B: Multiple Ascending Dose (Experimental): Participants will be randomized to receive multiple doses of VX-407.
  Interventions: Drug: VX-407
- Placebo Part B (Placebo Comparator): Participants will be randomized to receive placebo matched to VX-407.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VX-407 — Suspension for oral administration.
  Arms: Part A: Single Ascending Dose; Part B: Multiple Ascending Dose
Drug: Placebo — Suspension for oral administration.
  Arms: Placebo Part A; Placebo Part B

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability and pharmacokinetics of VX-407 in healthy participants.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4) (A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 32.0 kilogram per meter square (kg/m^2)
* A total body weight of greater than (>) 50 kg
* Nonsmoker or ex-smoker for at least 3 months before screening

Key Exclusion Criteria:

* History of febrile illness or other acute illness that has not fully resolved within 14 days before the first dose of study drug
* Any condition possibly affecting drug absorption

Other protocol defined Inclusion/Exclusion criteria will apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2026-03-03 (Estimated); Study Completion 2026-03-03 (Estimated)

PRIMARY OUTCOMES:
Part A: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Enrollment up to Day 10
Part B: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Enrollment up to Day 23

SECONDARY OUTCOMES:
Part A: Maximum Observed Concentration (Cmax) of VX-407 in Plasma | From Day 1 up to Day 6
Part B: Cmax of VX-407 in Plasma | Days 1, 7, and 14 up to Day 19
Part A: Area Under the Concentration Versus Time Curve From the Time of Dosing Extrapolated to Infinity (AUC0-inf) of VX-407 in Plasma | From Day 1 up to Day 6
Part B: Area Under the Concentration Time-curve From 0 to 24 Hours (AUC0-24hr) of VX-407 in Plasma | Days 1, 7, and 14 up to Day 19
Part A: Time Taken for VX-407 to Reach Maximum Concentration (tmax) | From Day 1 up to Day 6
Part B: Time Taken for VX-407 to Reach Maximum Concentration (tmax) | Days 1, 7, and 14 up to Day 19
Part A: Renal Clearance (CLr) of VX-407 | From Day 1 up to Day 6
Part B: CLr of VX-407 | Day 1 and Day 14

CONTACTS AND LOCATIONS:
Locations (1):
- ICON Lenexa, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/our-science/clinical-trials-data-sharing/